CLINICAL TRIAL: NCT02597413
Title: Evaluation of Post-voiding Residual Urine: a Before-after, Post-partum Study
Acronym: RPM-Eval
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/MN-01
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Postpartum Women
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before group: Women in this group are included before the implementation of a strategy of systematic catheterization (they will not be catheterized).
- After group: Women in this group are included after the implementation of a department-wide strategy of systematic catheterization.
  Intervention: catheterization
  Interventions: Procedure: Catheterization

INTERVENTIONS:
Procedure: Catheterization — Women in this group will be systematically catheterized before leaving the delivery room.
  Groups: After group

SUMMARY:
The primary objective of this study is to evaluate the impact of systematic catheter-drainage of urine for parturient women immediately in the delivery room on the occurrence of post-voiding urine residue.

DETAILED DESCRIPTION:
Secondarily, we will evaluate the impact of systematic catheter-drainage of urine for parturient women immediately in the delivery room on the occurrence of acute urine retention (first voiding volume > 500cc) and on post-partum bacteriuria rates.

ELIGIBILITY:
Inclusion Criteria:

* Paturient women admitted to the delivery room

Exclusion Criteria:

* Patients who have been catheterized during the third trimester of the current pregnancy
* History of surgery on the urinary tract

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all paturient women admitted to delivery rooms.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a post-voiding residue | Day 0 to Day 2 (just after first voiding)
  Assessed just after the first post-partum voiding.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Neron, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France